CLINICAL TRIAL: NCT04318548
Title: A Phase IIIB, Randomized, Observer-blind, Multicenter Study to Assess the Safety and Immunogenicity of GSK's Meningococcal Group B Vaccine When Administered Concomitantly With GSK's Meningococcal MenACWY Conjugate Vaccine to Healthy Subjects of 16-18 Years of Age
Brief Title: Study to Assess the Safety and Immunogenicity of GSK Meningococcal Group B Vaccine When Administered Concomitantly With GSK Meningococcal MenACWY Conjugate Vaccine in Healthy Subjects of 16-18 Years of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 205419; 2016-003722-16 (EudraCT Number)
Record Dates: First submitted 2020-03-20; First posted 2020-03-24 (Actual); Results first posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Infections, Meningococcal
Keywords: Meningitis; Invasive meningococcal disease; Bexsero; Menveo
MeSH Terms: conditions — Meningococcal Infections; Meningitis | interventions — 4CMenB vaccine; Meningococcal Vaccines; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is an Observer-blinded study. Recipients & study evaluators were unaware of vaccine administered.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- MenB+MenACWY Group (Experimental): Participants received 1 dose of rMenB+OMV NZ vaccine administered concomitantly with 1 dose of MenACWY vaccine, as separate injections in each arm at Day 1, 1 dose of rMenB+OMV NZ vaccine at Day 61 and 1 dose of placebo at Day 91.
  Interventions: Combination Product: Meningococcal Group B Vaccine (GSK3536829A) (rMenB+OMV NZ); Biological: Meningococcal MenACWY Conjugate Vaccine (GSK3536820A) (MenA lyo + MenCWY liquid); Combination Product: Placebo
- MenB Group (Experimental): Participants received 1 dose of rMenB+OMV NZ vaccine administered concomitantly with 1 dose of placebo, as separate injections in each arm at Day 1, 1 dose of rMenB+OMV NZ vaccine at Day 61 and 1 dose of MenACWY at Day 91.
  Interventions: Combination Product: Meningococcal Group B Vaccine (GSK3536829A) (rMenB+OMV NZ); Biological: Meningococcal MenACWY Conjugate Vaccine (GSK3536820A) (MenA lyo + MenCWY liquid); Combination Product: Placebo
- MenACWY Group (Experimental): Participants received 1 dose of MenACWY vaccine administered concomitantly with 1 dose of placebo, as separate injections in each arm at Day1, 1 dose of rMenB+OMV NZ vaccine each administered at Day 61 and at Day 91.
  Interventions: Combination Product: Meningococcal Group B Vaccine (GSK3536829A) (rMenB+OMV NZ); Biological: Meningococcal MenACWY Conjugate Vaccine (GSK3536820A) (MenA lyo + MenCWY liquid); Combination Product: Placebo

INTERVENTIONS:
Combination Product: Meningococcal Group B Vaccine (GSK3536829A) (rMenB+OMV NZ) — 1 dose of rMenB+OMV administered intramuscularly at day 1 and 61 to participants in MenB+MenACWY group and MenB group and as 1 dose at day 91 to participants in MenACWY group.
  Other Names: Bexsero
Biological: Meningococcal MenACWY Conjugate Vaccine (GSK3536820A) (MenA lyo + MenCWY liquid) — 1 dose of MenACWY administered intramuscularly at day 1 to participants in MenB+MenACWY group and MenACWY group, 1 dose at day 91 to participants for MenB group.
  Other Names: Menveo
Combination Product: Placebo — 1 dose of Placebo administered intramuscularly at 1 to participants in MenB group and MenACWY group and as 1 dose at day 91 to participants in MenB+MenACWY group.
  Other Names: NaCl, saline solution

SUMMARY:
The purpose of this study is to evaluate the immunogenicity, safety and tolerability of rMenB+OMV NZ and MenACWY vaccines when concomitantly administered to healthy subjects 16-18 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Participants who, in the opinion of the investigator, can and will comply with the requirements of the protocol or/and participants' parent(s)/Legally Acceptable Representative(s) [LAR(s)] who, in the opinion of the investigator, can and will comply, with the requirements of the protocol.
* Previous vaccination with 1 dose of quadrivalent meningococcal conjugate vaccine (MenACWY, Menveo or Menactra) at least 4 years prior to informed consent and assent as applicable.
* Written or /witnessed/thumb printed informed consent obtained from the participant/parent(s)/LAR(s) of the participant prior to performance of any study specific procedure.
* Written informed assent obtained from the participant (if applicable) along with informed consent from the participant's parent(s)/LAR(s) prior to performing any study specific procedure.
* A male or female between, and including, 16 and 18 years of age at the time of the first vaccination.
* Healthy participants as established by medical history and clinical examination before entering the study.
* Female participants of non-childbearing potential may be enrolled in the study. Non-childbearing potential is defined as pre-menarche, current bilateral tubal ligation or occlusion, hysterectomy, bilateral ovariectomy or post-menopause.
* Female participants of childbearing potential may be enrolled in the study if the participant:

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination, and
  * has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series.

Exclusion Criteria:

Medical conditions

* Progressive, unstable, or uncontrolled clinical conditions.
* Clinical conditions representing a contraindication to intramuscular vaccination and blood draws.
* Abnormal function of the immune system resulting from:

  * Clinical conditions.
  * Systemic administration of corticosteroids (PO/IV/IM) for more than 14 consecutive days within 90 days prior to study vaccination. This will mean prednisone ≥ 20 mg/day (for adult participants) or ≥ 0.5 mg/kg/day or 20 mg/day whichever is the maximum dose for pediatric participants, or equivalent. Inhaled and topical steroids are allowed.
  * Administration of antineoplastic or immunomodulating agents or radiotherapy within 90 days prior to informed consent.
* Any other clinical condition that, in the opinion of the investigator, might pose additional risk to the participant due to participation in the study.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccines.
* History of any reaction or hypersensitivity likely to be exacerbated by any medicinal products or medical equipment whose use is foreseen in this study.
* Current or previous, confirmed, or suspected disease caused by N. meningitidis.
* Known contact to an individual with any laboratory-confirmed N. meningitidis infection within 60 days, prior to enrolment.
* History of neuroinflammatory or autoimmune condition.
* Recurrent history or un-controlled neurological disorders or seizures.

Prior/Concomitant therapy

* Use of any investigational or non-registered product other than the study vaccine(s) during the period starting 30 days before the informed consent or planned use during the study period.
* Administration of immunoglobulins and/or any blood products or plasma derivatives during the period starting 180 days before the informed consent or planned administration during the study period.
* Previous vaccination with any group B meningococcal vaccine at any time prior to informed consent and assent as applicable.
* Previous vaccination with 2 doses of quadrivalent meningococcal conjugate vaccine (MenACWY, Menveo, Menactra or MenQuadfi).

Prior/Concurrent clinical study experience

• Participant concurrently participating in another clinical study, at any time during the study period, in which the participant has been or will be exposed to an investigational or a non-investigational vaccine/product, will not be enrolled.

Other exclusions

* Child in care.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.
* Any study personnel or immediate dependents, family, or household member.

Ages: 16 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 945 (Actual)
Dates: Start 2020-08-25 (Actual); Primary Completion 2023-11-21 (Actual); Study Completion 2023-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (41):
- United States (38):
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Bell Gardens, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Oakland, California
  - GSK Investigational Site, Roseville, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, San Jose, California
  - GSK Investigational Site, Santa Clara, California
  - GSK Investigational Site, Walnut Creek, California
  - GSK Investigational Site, Wellington, Florida
  - GSK Investigational Site, Boise, Idaho
  - GSK Investigational Site, Nampa, Idaho
  - GSK Investigational Site, Evansville, Indiana
  - GSK Investigational Site, Bardstown, Kentucky
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Lafayette, Louisiana
  - GSK Investigational Site, Lincoln, Nebraska
  - GSK Investigational Site, Cortland, New York
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Corvallis, Oregon
  - GSK Investigational Site, Erie, Pennsylvania
  - GSK Investigational Site, Hermitage, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Sioux Falls, South Dakota
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Plano, Texas
  - GSK Investigational Site, Victoria, Texas
  - GSK Investigational Site, Waxahachie, Texas
  - GSK Investigational Site, Orem, Utah
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, South Jordan, Utah
  - GSK Investigational Site, Syracuse, Utah
  - GSK Investigational Site, Falls Church, Virginia
  - GSK Investigational Site, Richmond, Virginia
- Italy (3):
  - GSK Investigational Site, Chiavari GE
  - GSK Investigational Site, Foggia
  - GSK Investigational Site, Milan

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study ended on Day 271 for participants who had not reached Day 271 when Protocol Amendment 7 took effect, and on Day 451 for those who had already passed Day 271.
  Safety follow-up period for each participant was from Day 1 up to Day 451 or Day 271 for participants who have not reached Day 271 at the time Protocol Amendment 7 took effect.
Pre-assignment Details: Out of 945 participants enrolled, only 940 were randomized into the three treatment groups. After randomization, two participants did not receive the vaccination, so only 938 participants were included in the Exposed Set and started the study.
Period: Overall Study
Arm/Group | MenB+MenACWY Group | MenB Group | MenACWY Group
Started | 310 | 308 | 320
Completed | 297 | 284 | 298
Not Completed | 13 | 24 | 22
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Lost to Follow-up | 6 | 13 | 9
Not completed — Protocol Violation | 1 | 0 | 2
Not completed — Consent withdrawal, not due to a (S)AE | 5 | 9 | 6
Not completed — Migrated / moved from the study area | 0 | 0 | 1
Not completed — Other | 1 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MenB+MenACWY Group | MenB Group | MenACWY Group | Total
Number analyzed (Participants) | 310 | 308 | 320 | 938
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.4 (0.7) | 16.4 (0.7) | 16.5 (0.7) | 16.4 (0.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 156 | 138 | 163 | 457
  Male | 154 | 170 | 157 | 481
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 46 | 38 | 37 | 121
  Not Hispanic or Latino | 263 | 270 | 282 | 815
  Unknown or Not Reported | 1 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Solicited Local Adverse Events (AEs) After the Vaccination With rMenB+OMV NZ
Description: Solicited local adverse events assessed are injection site pain, erythema, swelling, induration. Any solicited local AEs = occurrence of the symptom regardless of intensity grade.
Time Frame: During 7 days after the rMenB+OMV NZ vaccination at Day 1
Population: Analysis was performed on the Exposed set (ES), which included all participants who received at least one dose of the study treatment and had the electronic diary (eDiary) for solicited events completed after the administration of study treatment and for whom data were available during the specified period. Allocation per group is based on the treatment administered. Only participants with data available at specified timepoints were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | MenB+MenACWY Group | MenB Group | MenACWY Group
Number analyzed (Participants) | 307 | 306 | 0
Participants
  Erythema | 12 | 12 |
  Induration | 14 | 22 |
  Pain | 246 | 247 |
  Swelling | 15 | 18 |

2. Primary Outcome: Number of Participants With Solicited Local Adverse Events (AEs) After the Vaccination With rMenB+OMV NZ
Description: as for outcome 1
Time Frame: During 7 days after the rMenB+OMV NZ vaccination at Day 61
Population: Analysis was performed on the Exposed set (ES), which included all participants who received at least one dose of the study treatment and had the eDiary for solicited events completed after the administration of study treatment and for whom data were available during the specified period. Allocation per group is based on the treatment administered.
Measure: Count of Participants; unit: Participants
Arm/Group | MenB+MenACWY Group | MenB Group | MenACWY Group
Number analyzed (Participants) | 283 | 269 | 287
Participants
  Erythema: number analyzed (Participants) | 283 | 268 | 287
  Erythema | 17 | 17 | 8
  Induration: number analyzed (Participants) | 283 | 268 | 287
  Induration | 18 | 19 | 6
  Pain | 240 | 228 | 238
  Swelling: number analyzed (Participants) | 283 | 268 | 287
  Swelling | 16 | 16 | 7

3. Primary Outcome: Number of Participants With Solicited Local Adverse Events (AEs) After the Vaccination With rMenB+OMV NZ
Description: as for outcome 1
Time Frame: During 7 days after the rMenB+OMV NZ vaccination at Day 91
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | MenB+MenACWY Group | MenB Group | MenACWY Group
Number analyzed (Participants) | 0 | 0 | 269
Participants
  Erythema |  |  | 14
  Induration |  |  | 11
  Pain |  |  | 205
  Swelling |  |  | 13

4. Primary Outcome: Number of Participants With Solicited Local AEs After the Vaccination With MenACWY
Description: Solicited local adverse events assessed are injection site pain, erythema, swelling, induration. Any solicited local AEs= occurrence of the symptom regardless of intensity grade.
Time Frame: During 7 days after the MenACWY vaccination at Day 1
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | MenB+MenACWY Group | MenB Group | MenACWY Group
Number analyzed (Participants) | 307 | 0 | 319
Participants
  Erythema | 5 |  | 6
  Induration | 7 |  | 7
  Pain | 93 |  | 104
  Swelling | 5 |  | 5

5. Primary Outcome: Number of Participants With Solicited Local AEs After the Vaccination With MenACWY
Description: as for outcome 4
Time Frame: During 7 days after the MenACWY vaccination at Day 61
Population: Analysis was performed on the ES, which included all participants who received at least one dose of the study treatment and had the eDiary for solicited events completed after the administration of study treatment and for whom data were available during the specified period. Allocation per group is based on the treatment administered. 1 participant in MenB Group received wrong study treatment at Day 61 (MenACWY vaccine instead of rMenB+OMV NZ), hence was considered in the analysis population.
Measure: Count of Participants; unit: Participants
Arm/Group | MenB+MenACWY Group | MenB Group | MenACWY Group
Number analyzed (Participants) | 0 | 1 | 0
Participants
  Erythema |  | 0 |
  Induration |  | 0 |
  Pain |  | 1 |
  Swelling |  | 0 |

6. Primary Outcome: Number of Participants With Solicited Local AEs After the Vaccination With MenACWY
Description: as for outcome 4
Time Frame: During 7 days after the MenACWY vaccination at Day 91
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | MenB+MenACWY Group | MenB Group | MenACWY Group
Number analyzed (Participants) | 0 | 265 | 0
Participants
  Erythema: number analyzed (Participants) | 0 | 264 | 0
  Erythema |  | 4 |
  Induration: number analyzed (Participants) | 0 | 263 | 0
  Induration |  | 1 |
  Pain: number analyzed (Participants) | 0 | 264 | 0
  Pain |  | 38 |
  Swelling |  | 5 |

7. Primary Outcome: Number of Participants With Solicited Local AEs After the Vaccination With Placebo
Description: as for outcome 1
Time Frame: During 7 days after the Placebo vaccination at Day 1
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | MenB+MenACWY Group | MenB Group | MenACWY Group
Number analyzed (Participants) | 0 | 306 | 320
Participants
  Erythema |  | 2 | 2
  Induration |  | 5 | 0
  Pain |  | 78 | 77
  Swelling |  | 2 | 1

8. Primary Outcome: Number of Participants With Solicited Local AEs After the Vaccination With Placebo
Description: as for outcome 1
Time Frame: During 7 days after the Placebo vaccination at Day 91
Population: Analysis was performed on the ES, which included all participants who received at least one dose of the study treatment and had the eDiary for solicited events completed after the administration of study treatment and for whom data were available during the specified period. Allocation per group is based on the treatment administered. 1 participant in MenACWY Group received wrong study treatment at Day 91 (placebo instead of rMenB+OMV NZ), hence was considered in the analysis population.
Measure: Count of Participants; unit: Participants
Arm/Group | MenB+MenACWY Group | MenB Group | MenACWY Group
Number analyzed (Participants) | 282 | 0 | 1
Participants
  Erythema | 1 |  | 0
  Induration | 1 |  | 0
  Pain | 25 |  | 0
  Swelling | 0 |  | 0

9. Primary Outcome: Number of Participants With Solicited Systemic AEs
Description: Solicited systemic adverse events assessed are fever [temperature >= 38.0°C], nausea, fatigue, myalgia, arthralgia, and headache.
Time Frame: During 7 days after the first study intervention administration occurring at Day 1
Population: Analysis was performed on the Exposed set (ES), which included all participants who received at least one dose of the study treatment and had the eDiary for solicited events completed after the administration of study treatment and for whom data were available during the specified period.
Measure: Count of Participants; unit: Participants
Arm/Group | MenB+MenACWY Group | MenB Group | MenACWY Group
Number analyzed (Participants) | 307 | 306 | 320
Participants
  Arthralgia | 24 | 32 | 24
  Fatigue | 114 | 118 | 108
  Headache | 128 | 135 | 134
  Myalgia | 36 | 49 | 31
  Nausea | 46 | 57 | 51
  Fever | 7 | 10 | 2

10. Primary Outcome: Number of Participants With Solicited Systemic AEs
Description: as for outcome 9
Time Frame: During 7 days after the second study intervention administration occurring at Day 61
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | MenB+MenACWY Group | MenB Group | MenACWY Group
Number analyzed (Participants) | 284 | 269 | 287
Participants
  Arthralgia: number analyzed (Participants) | 283 | 269 | 287
  Arthralgia | 28 | 24 | 27
  Fatigue: number analyzed (Participants) | 283 | 269 | 287
  Fatigue | 96 | 101 | 88
  Headache: number analyzed (Participants) | 283 | 269 | 287
  Headache | 112 | 103 | 93
  Myalgia: number analyzed (Participants) | 283 | 269 | 287
  Myalgia | 41 | 42 | 43
  Nausea: number analyzed (Participants) | 283 | 269 | 287
  Nausea | 37 | 37 | 40
  Fever | 4 | 8 | 6

11. Primary Outcome: Number of Participants With Solicited Systemic AEs
Description: as for outcome 9
Time Frame: During 7 days after the third study intervention administration occurring at Day 91
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | MenB+MenACWY Group | MenB Group | MenACWY Group
Number analyzed (Participants) | 282 | 263 | 270
Participants
  Arthralgia | 7 | 8 | 24
  Fatigue | 38 | 59 | 86
  Headache | 56 | 53 | 84
  Myalgia | 7 | 16 | 39
  Nausea | 20 | 18 | 31
  Fever | 2 | 2 | 6

12. Primary Outcome: Number of Participants With Any Unsolicited AEs (Including All Serious Adverse Events)
Description: Unsolicited adverse events are defined as any AE reported in addition to those solicited during the clinical study. Also, any 'solicited' symptom with onset outside the specified period of follow-up for solicited symptoms are reported as an unsolicited adverse event. Any solicited AE that has not resolved within 30 days post vaccination and is reported during clinic visits or safety follow-up calls is entered into the subject's electronic Case Report Form (eCRF) as an unsolicited AE. Serious Adverse Events (SAEs) are any untoward medical occurrence that result in death, are life-threatening, require hospitalization or prolongation of existing hospitalization, result in disability/incapacity and is a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: During 30 days after the first study intervention administration occurring at Day 1
Population: Analysis was performed on the Exposed set (ES). Only participants with data available at specified timepoints were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | MenB+MenACWY Group | MenB Group | MenACWY Group
Number analyzed (Participants) | 310 | 308 | 320
Participants | 49 | 54 | 55

13. Primary Outcome: Number of Participants With Any Unsolicited AEs (Including All Serious Adverse Events)
Description: as for outcome 12
Time Frame: During 30 days after the second study intervention administration occurring at Day 61
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | MenB+MenACWY Group | MenB Group | MenACWY Group
Number analyzed (Participants) | 310 | 308 | 320
Participants | 51 | 47 | 44

14. Primary Outcome: Number of Participants With Any Unsolicited AEs (Including All Serious Adverse Events)
Description: as for outcome 12
Time Frame: During 30 days after the third study intervention administration occurring at Day 91
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | MenB+MenACWY Group | MenB Group | MenACWY Group
Number analyzed (Participants) | 310 | 308 | 320
Participants | 37 | 37 | 38

15. Primary Outcome: Number of Participants With Any AEs/SAEs Leading to Withdrawal
Description: Unsolicited AEs are defined as any AE reported in addition to those solicited during the clinical study. Also, any 'solicited' symptom with onset outside the specified period of follow-up for solicited symptoms are reported as an unsolicited adverse event. Any solicited AE that has not resolved within 30 days post vaccination and is reported during clinic visits or safety follow-up calls is entered into the subject's electronic Case Report Form (eCRF) as an unsolicited AE. SAEs are any untoward medical occurrence that result in death, are life-threatening, require hospitalization or prolongation of existing hospitalization, result in disability/incapacity and is a congenital anomaly/birth defect in the offspring of a study subject. A participant was considered a 'withdrawal' from the study when no study procedure has occurred, no follow-up has been performed and no further information has been collected for this participant from the date of withdrawal/last contact.
Time Frame: During 30 days after the first study intervention administration occurring at Day 1
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | MenB+MenACWY Group | MenB Group | MenACWY Group
Number analyzed (Participants) | 310 | 308 | 320
Participants | 0 | 0 | 1

16. Primary Outcome: Number of Participants With Any AEs/SAEs Leading to Withdrawal
Description: as for outcome 15
Time Frame: During 30 days after the second study intervention administration occurring at Day 61
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | MenB+MenACWY Group | MenB Group | MenACWY Group
Number analyzed (Participants) | 310 | 308 | 320
Participants | 0 | 0 | 0

17. Primary Outcome: Number of Participants With Any AEs/SAEs Leading to Withdrawal
Description: as for outcome 15
Time Frame: During 30 days after the third study intervention administration occurring at Day 91
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | MenB+MenACWY Group | MenB Group | MenACWY Group
Number analyzed (Participants) | 310 | 308 | 320
Participants | 0 | 0 | 0

18. Primary Outcome: Number of Participants With Any Medically Attended AEs
Description: Medically attended AEs are symptoms or illnesses requiring hospitalization, or emergency room visit, or visit to/by a health care provider.
Time Frame: During 30 days after the first study intervention administration occurring at Day 1
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | MenB+MenACWY Group | MenB Group | MenACWY Group
Number analyzed (Participants) | 310 | 308 | 320
Participants | 28 | 36 | 26

19. Primary Outcome: Number of Participants With Any Medically Attended AEs
Description: as for outcome 18
Time Frame: During 30 days after the second study intervention administration occurring at Day 61
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | MenB+MenACWY Group | MenB Group | MenACWY Group
Number analyzed (Participants) | 310 | 308 | 320
Participants | 28 | 32 | 25

20. Primary Outcome: Number of Participants With Any Medically Attended AEs
Description: as for outcome 18
Time Frame: During 30 days after the third study intervention administration occurring at Day 91
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | MenB+MenACWY Group | MenB Group | MenACWY Group
Number analyzed (Participants) | 310 | 308 | 320
Participants | 19 | 21 | 17

21. Primary Outcome: Number of Participants With Any SAEs, AEs Leading to Withdrawal and Medically Attended AEs
Description: SAEs, AEs leading to withdrawal and medically attended AEs were assessed throughout the study period are reported in this outcome measure.
Time Frame: Throughout the study period (Day 1 to Day 271)
Population: Analysis was performed on the Exposed set (ES), which included all participants who received at least one dose of the study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | MenB+MenACWY Group | MenB Group | MenACWY Group
Number analyzed (Participants) | 310 | 308 | 320
Participants
  SAEs | 2 | 3 | 5
  AEs leading to withdrawal | 0 | 0 | 1
  Medically attended AEs | 93 | 103 | 96

22. Primary Outcome: Number of Participants Who Received rMenB+OMV NZ With Adverse Events of Special Interest (AESI)
Description: AESIs are predefined (serious or non-serious) adverse events of scientific and medical concern specific to the product or program, for which ongoing monitoring and rapid communication by the investigator to the sponsor can be appropriate, because such an event might warrant further investigation in order to characterize and understand it.
Time Frame: Throughout the study period (Day 1 to Day 271)
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | MenB+MenACWY Group | MenB Group | MenACWY Group
Number analyzed (Participants) | 310 | 308 | 320
Participants | 0 | 0 | 0

23. Primary Outcome: Number of Participants With Any SAEs and AEs Leading to Withdrawal
Description: as for outcome 15
Time Frame: During safety follow-up (Day 271 to Day 451)
Population: Analysis was performed on the Exposed set (ES). Only participants with data available at specified timepoints (during safety follow-up period from Day 271 to Day 451) were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | MenB+MenACWY Group | MenB Group | MenACWY Group
Number analyzed (Participants) | 88 | 90 | 87
Participants
  SAEs | 0 | 1 | 2
  AEs leading to withdrawal | 0 | 0 | 0

24. Primary Outcome: Number of Participants Who Received rMenB+OMV NZ With AESI
Description: as for outcome 22
Time Frame: During safety follow-up (Day 271 to Day 451)
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | MenB+MenACWY Group | MenB Group | MenACWY Group
Number analyzed (Participants) | 88 | 90 | 87
Participants | 0 | 0 | 0

25. Primary Outcome: Human Serum Bactericidal Assay (hSBA) Geometric Mean Titers (GMTs) Against Each of the N. Meningitidis Serogroup B Strains at 1 Month After the Second Vaccination With rMenB+OMV NZ (Groups MenB+MenACWY and MenB), and Between-group GMT Ratios
Description: hSBA titers were measured by serum bactericidal assay and expressed as Geometric Mean Titers (GMTs) against N. meningitidis serogroup B indicator strains (M14459 [fHbp], 96217 [NadA], NZ98/254 [PorA] and M13520 [NHBA]).
Time Frame: At Day 91 (1 month after the second vaccination with rMenB+OMV NZ in MenB+MenACWY and MenB groups)
Population: Analysis was performed on the Per Protocol Set (PPS), which included participants who received at least 1 dose of the study intervention to which they were randomized and had post-vaccination data available at the specified timepoint minus participants with protocol deviations that led to exclusion from the PPS.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | MenB+MenACWY Group | MenB Group
Number analyzed (Participants) | 274 | 267
Titers
  fHbp (M14459): number analyzed (Participants) | 274 | 266
  fHbp (M14459) | 16.9 [14.4 to 19.8] | 18.7 [15.9 to 21.9]
  NadA (96217) | 239.6 [202.9 to 283.0] | 272.4 [231.1 to 321.0]
  PorA (NZ98/254): number analyzed (Participants) | 273 | 266
  PorA (NZ98/254) | 18.8 [15.6 to 22.6] | 21.3 [17.7 to 25.6]
  NHBA (M13520): number analyzed (Participants) | 273 | 266
  NHBA (M13520) | 19.0 [15.6 to 23.1] | 20.5 [16.9 to 24.9]
Statistical Analysis 1: Comparison: MenB+MenACWY Group vs MenB Group; To demonstrate the non-inferiority (NI) of the antibody response to rMenB+OMV NZ given concomitantly with MenACWY compared to rMenB+OMV NZ administered alone, measured by hSBA GMTs against N. meningitidis serogroup B indicator strains at one month after the second vaccination with rMenB+OMV NZ (at Day 91); Test type: Non-Inferiority — NI was to be demonstrated if the lower limit (LL) of the 2-sided 95% CI of the GMT ratio between the MenB+MenACWY group and MenB group for hSBA titers against M14459 (fHbp) strain was above (>) 0.5; ANOVA; GMT Ratio = 0.90, 95% CI 2-sided [0.77 to 1.06] — The ratio of GMTs (MenB+MenACWY/MenB) and the corresponding CI is constructed by exponentiating the mean difference and the confidence limits in log10 (titer), using ANOVA with study centre included as an independent variable
Statistical Analysis 2: Comparison: MenB+MenACWY Group vs MenB Group; To demonstrate the non-inferiority of the antibody response to rMenB+OMV NZ given concomitantly with MenACWY compared to rMenB+OMV NZ administered alone, measured by hSBA GMTs against N. meningitidis serogroup B indicator strains at one month after the second vaccination with rMenB+OMV NZ (at Day 91); Test type: Non-Inferiority — NI was to be demonstrated if LL of the 2-sided 95% CI of the GMT ratio between the MenB+MenACWY group and MenB group for hSBA titers against 96217 (NadA) strain was >0.5; ANOVA; GMT Ratio = 0.88, 95% CI 2-sided [0.75 to 1.04] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 3: Comparison: MenB+MenACWY Group vs MenB Group; [analysis description as in outcome 25, analysis 2]; Test type: Non-Inferiority — NI was to be demonstrated if LL of the 2-sided 95% CI of the GMT ratio between the MenB+MenACWY group and MenB group for hSBA titers against NZ98/254 (PorA) strain was >0.5; ANOVA; GMT Ratio = 0.93, 95% CI 2-sided [0.76 to 1.12] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 4: Comparison: MenB+MenACWY Group vs MenB Group; [analysis description as in outcome 25, analysis 2]; Test type: Non-Inferiority — NI was to be demonstrated if LL of the 2-sided 95% CI of the GMT ratio between the MenB+MenACWY group and MenB group for hSBA titers against M13520 (NHBA) strain was >0.5; ANOVA; GMT Ratio = 0.88, 95% CI 2-sided [0.73 to 1.06] — [estimate comment as in outcome 25, analysis 1]

26. Primary Outcome: hSBA GMTs Against Each of the N. Meningitidis Serogroups A, C, W and Y After Vaccination With MenACWY (Groups MenB+MenACWY and MenACWY), and Between-group GMT Ratios
Description: hSBA titers were measured by serum bactericidal assay and expressed as GMTs against each of the 4 serogroups Men A, Men C, Men W and Men Y.
Time Frame: At Day 31 (1 month after the vaccination with MenACWY in MenACWY and MenB+MenACWY groups)
Population: Analysis was performed on the Per Protocol Set (PPS). Only those participants with data available at specified timepoint were included in analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | MenB+MenACWY Group | MenACWY Group
Number analyzed (Participants) | 295 | 303
Titers
  Men A: number analyzed (Participants) | 290 | 292
  Men A | 2388.8 [1977.2 to 2886.1] | 2536.1 [2095.7 to 3069.1]
  Men C: number analyzed (Participants) | 295 | 302
  Men C | 2075.9 [1602.5 to 2689.3] | 1867.6 [1438.7 to 2424.2]
  Men W | 2299.3 [1902.5 to 2778.9] | 2305.7 [1905.3 to 2790.4]
  Men Y | 2897.3 [2359.2 to 3558.3] | 2802.0 [2278.3 to 3446.2]
Statistical Analysis 1: Comparison: MenB+MenACWY Group vs MenACWY Group; To demonstrate the non-inferiority of the antibody response to MenACWY given concomitantly with rMenB+OMV NZ compared to MenACWY administered alone, as measured by hSBA GMTs against the N. meningitidis serogroup Men A, at one month after the vaccination with MenACWY (at Day 31); Test type: Non-Inferiority — NI was to be demonstrated if LL of the 2-sided 95% CI of the between-group ratio of hSBA GMTs between MenB+MenACWY group and MenACWY group for Men A serogroup was >0.5; ANOVA; GMT Ratio = 0.94, 95% CI 2-sided [0.78 to 1.14] — The ratio of GMTs (MenB+MenACWY/MenACWY) and the corresponding CI is constructed by exponentiating the mean difference and the confidence limits in log10 (titer), using ANOVA with study centre included as an independent variable
Statistical Analysis 2: Comparison: MenB+MenACWY Group vs MenACWY Group; To demonstrate the non-inferiority of the antibody response to MenACWY given concomitantly with rMenB+OMV NZ compared to MenACWY administered alone, as measured by hSBA GMTs against the N. meningitidis serogroup Men C, at one month after the vaccination with MenACWY (at Day 31); Test type: Non-Inferiority — NI was to be demonstrated if LL of the 2-sided 95% CI of the between-group ratio of hSBA GMTs between MenB+MenACWY group and MenACWY group for Men C serogroup was >0.5; ANOVA; GMT Ratio = 1.11, 95% CI 2-sided [0.86 to 1.44] — [estimate comment as in outcome 26, analysis 1]
Statistical Analysis 3: Comparison: MenB+MenACWY Group vs MenACWY Group; To demonstrate the non-inferiority of the antibody response to MenACWY given concomitantly with rMenB+OMV NZ compared to MenACWY administered alone, as measured by hSBA GMTs against the N. meningitidis serogroup Men W, at one month after the vaccination with MenACWY (at Day 31); Test type: Non-Inferiority — NI was to be demonstrated if LL of the 2-sided 95% CI of the between-group ratio of hSBA GMTs between MenB+MenACWY group and MenACWY group for Men W serogroup was >0.5; ANOVA; GMT Ratio = 1.00, 95% CI 2-sided [0.82 to 1.21] — [estimate comment as in outcome 26, analysis 1]
Statistical Analysis 4: Comparison: MenB+MenACWY Group vs MenACWY Group; To demonstrate the non-inferiority of the antibody response to MenACWY given concomitantly with rMenB+OMV NZ compared to MenACWY administered alone, as measured by hSBA GMTs against the N. meningitidis serogroup Men Y, at one month after the vaccination with MenACWY (at Day 31); Test type: Non-Inferiority — NI was to be demonstrated if LL of the 2-sided 95% CI of the between-group ratio of hSBA GMTs between MenB+MenACWY group and MenACWY group for Men Y serogroup was >0.5; ANOVA; GMT Ratio = 1.03, 95% CI 2-sided [0.84 to 1.27] — [estimate comment as in outcome 26, analysis 1]

27. Secondary Outcome: hSBA Geometric Mean Concentrations (GMCs) Measured by ECL Against Each of the N. Meningitidis Serogroups After MenACWY Vaccination
Description: Immune response to MenACWY given with or without rMenB+OMV NZ, as measured by ectrochemiluminescence-based multiplex (ECL) GMCs against each of the serogroups A, C, W and Y. ECL (validated assay) was used because ELISA is not validated.
Time Frame: At Day 31 (1 month after the vaccination of MenACWY in MenACWY and MenB+MenACWY groups)
Reporting Status: Not Posted

28. Secondary Outcome: hSBA GMTs Against Each of the Serogroup B Strains in Both MenB+MenACWY and MenB Groups After First rMenB+OMV NZ Vaccination and Between-group GMT Ratios
Description: hSBA titers were measured by bactericidal activity against N. meningitidis serogroup B indicator strains (M14459 [fHbp], 96217 [NadA], NZ98/254 [PorA] and M13520 [NHBA]) and expressed in GMTs.
Time Frame: At Day 31 (1 month after first vaccination with rMenB+OMV NZ)
Population: as for outcome 26
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | MenB+MenACWY Group | MenB Group
Number analyzed (Participants) | 294 | 294
Titers
  fHbp (M14459) | 4.3 [3.6 to 5.1] | 5.6 [4.7 to 6.7]
  NadA (96217) | 45.2 [36.0 to 56.9] | 73.4 [58.5 to 91.9]
  PorA (NZ98/254): number analyzed (Participants) | 294 | 293
  PorA (NZ98/254) | 4.2 [3.5 to 5.0] | 5.6 [4.7 to 6.6]
  NHBA (M13520): number analyzed (Participants) | 294 | 293
  NHBA (M13520) | 6.4 [5.1 to 8.1] | 8.8 [7.0 to 11.1]
Statistical Analysis 1: Comparison: MenB+MenACWY Group vs MenB Group; To assess the immune response to rMenB+OMV NZ given concomitantly with MenACWY compared to rMenB+OMV NZ administered alone, measured by hSBA GMTs against N. meningitidis M14459 (fHbp) strain at one month after the fisrt vaccination with rMenB+OMV NZ (at Day 31); Test type: Other; ANOVA; GMT Ratio = 0.76, 95% CI 2-sided [0.64 to 0.91] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 2: Comparison: MenB+MenACWY Group vs MenB Group; To assess the immune response to rMenB+OMV NZ given concomitantly with MenACWY compared to rMenB+OMV NZ administered alone, measured by hSBA GMTs against N. meningitidis 96217 (NadA) strain at one month after the first vaccination with rMenB+OMV NZ (at Day 31); Test type: Other; ANOVA; GMT Ratio = 0.62, 95% CI 2-sided [0.49 to 0.77] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 3: Comparison: MenB+MenACWY Group vs MenB Group; To assess the immune response to rMenB+OMV NZ given concomitantly with MenACWY compared to rMenB+OMV NZ administered alone, measured by hSBA GMTs against N. meningitidis NZ98/254 (PorA) strain at one month after the first vaccination with rMenB+OMV NZ (at Day 31); Test type: Other; ANOVA; GMT Ratio = 0.73, 95% CI 2-sided [0.58 to 0.91] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 4: Comparison: MenB+MenACWY Group vs MenB Group; To assess the immune response to rMenB+OMV NZ given concomitantly with MenACWY compared to rMenB+OMV NZ administered alone, measured by hSBA GMTs against N. meningitidis M13520 (NHBA) at one month after the first vaccination with rMenB+OMV NZ (at Day 31); Test type: Other; ANOVA; GMT Ratio = 0.76, 95% CI 2-sided [0.64 to 0.90] — [estimate comment as in outcome 25, analysis 1]

29. Secondary Outcome: Geometric Mean Ratios (GMRs) Against Each of the N. Meningitidis Serogroup B Strains in Both MenB+MenACWY and MenB Groups After the First rMenB+OMV NZ Vaccination
Description: The immune response to rMenB+OMV NZ was measured by bactericidal activity against N. meningitidis serogroup B indicator strains (M14459 [fHbp], 96217 [NadA], NZ98/254 [PorA] and M13520 [NHBA]) in terms of GMRs (after vaccination/baseline).
Time Frame: At Dya 31 (1 month after first rMenB+OMV NZ vaccination) compared to the baseline (Day 1)
Population: as for outcome 26
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | MenB+MenACWY Group | MenB Group
Number analyzed (Participants) | 294 | 294
Ratio
  fHbp (M14459) | 1.6 [1.4 to 1.9] | 2.0 [1.7 to 2.4]
  NadA (96217) | 5.9 [4.7 to 7.4] | 9.3 [7.5 to 11.6]
  PorA (NZ98/254): number analyzed (Participants) | 294 | 293
  PorA (NZ98/254) | 1.4 [1.2 to 1.6] | 1.8 [1.5 to 2.1]
  NHBA (M13520): number analyzed (Participants) | 294 | 293
  NHBA (M13520) | 1.8 [1.5 to 2.2] | 2.3 [1.9 to 2.8]

30. Secondary Outcome: GMRs Against Each of the N. Meningitidis Serogroup B Strains in Both MenB+MenACWY and MenB Groups After the Second rMenB+OMV NZ Vaccination
Description: as for outcome 29
Time Frame: At Day 91 (1 month after the second rMenB+OMV NZ vaccination) compared to the baseline (Day 1)
Population: as for outcome 26
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | MenB+MenACWY Group | MenB Group
Number analyzed (Participants) | 274 | 267
Ratio
  fHbp (M14459): number analyzed (Participants) | 274 | 266
  fHbp (M14459) | 6.4 [5.5 to 7.5] | 7.0 [5.9 to 8.1]
  NadA (96217) | 30.7 [25.8 to 36.6] | 35.1 [29.5 to 41.7]
  PorA (NZ98/254): number analyzed (Participants) | 273 | 266
  PorA (NZ98/254) | 6.0 [5.0 to 7.2] | 6.9 [5.8 to 8.3]
  NHBA (M13520): number analyzed (Participants) | 273 | 266
  NHBA (M13520) | 5.2 [4.4 to 6.2] | 5.6 [4.7 to 6.6]

31. Secondary Outcome: Percentage of Participants With hSBA Titers >= Lower Limit of Quantitation (LLOQ) for Each and All Serogroup B Test Strains in Both MenB+MenACWY and MenB Groups After the First rMenB+OMV NZ Vaccination
Description: The immune response to rMenB+OMV NZ vaccine is evaluated by measuring bactericidal activity in terms of participants with hSBA titers >= LLOQ against N. meningitidis serogroup B test strains (M14459 [fHbp], 96217 [NadA], NZ98/254 [PorA] and M13520 [NHBA]).
Time Frame: At Day 31 (one month after the first rMenB+OMV NZ vaccination)
Population: as for outcome 26
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MenB+MenACWY Group | MenB Group
Number analyzed (Participants) | 294 | 294
Percentage of participants
  fHbp (M14459) | 32.3 [27.0 to 38.0] | 44.9 [39.1 to 50.8]
  NadA (96217) | 77.9 [72.7 to 82.5] | 85.7 [81.2 to 89.5]
  PorA ( NZ98/254): number analyzed (Participants) | 294 | 293
  PorA ( NZ98/254) | 21.1 [16.6 to 26.2] | 30.4 [25.2 to 36.0]
  NHBA (M13520): number analyzed (Participants) | 294 | 293
  NHBA (M13520) | 37.1 [31.5 to 42.9] | 44.4 [38.6 to 50.3]

32. Secondary Outcome: Percentage of Participants With hSBA Titers >= LLOQ for Each and All of the Serogroup B Test Strains in Both MenB+MenACWY and MenB Groups After the Second rMenB+OMV NZ Vaccination
Description: as for outcome 31
Time Frame: At Day 91 (1 month after the second rMenB+OMV NZ vaccination)
Population: as for outcome 26
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MenB+MenACWY Group | MenB Group
Number analyzed (Participants) | 274 | 267
Percentage of participants
  fHbp (M14459 ): number analyzed (Participants) | 274 | 266
  fHbp (M14459 ) | 92.3 [88.5 to 95.2] | 92.5 [88.6 to 95.3]
  NadA (96217) | 99.6 [98.0 to 100] | 99.6 [97.9 to 100]
  PorA (NZ98/254): number analyzed (Participants) | 273 | 266
  PorA (NZ98/254) | 83.2 [78.2 to 87.4] | 85.0 [80.1 to 89.0]
  NHBA (M13520): number analyzed (Participants) | 273 | 266
  NHBA (M13520) | 84.2 [79.4 to 88.4] | 90.2 [86.0 to 93.5]

33. Secondary Outcome: Percentage of Participants With 4-fold Increase in hSBA Titers Relative to Baseline in Both MenB+MenACWY and MenB Groups After the First rMenB+OMV NZ Vaccination
Description: The immune response to rMenB+OMV NZ vaccine is evaluated by measuring bactericidal activity against each of N. meningitidis serogroup B test strains (M14459 [fHbp], 96217 [NadA], NZ98/254 [PorA] and M13520 [NHBA]) in terms of the Four-fold increase defined as: - For a pre-vaccination titer < limit of detection (LOD), a post-vaccination titer of >= 4-fold the LOD or >= LLOQ, whichever is greater, - For a pre-vaccination titer >= LOD but <LLOQ, a post vaccination titer of at least 4-fold the LLOQ, - For a pre-vaccination titer >= LLOQ, a post vaccination titer of at least 4-fold the pre-vaccination titer.
Time Frame: At 1 month after the first rMenB+OMV NZ vaccination (i.e at Day 31) relative to baseline (i.e. Day 1)
Population: as for outcome 26
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MenB+MenACWY Group | MenB Group
Number analyzed (Participants) | 293 | 293
Percentage of participants
  fHbp (M14459): number analyzed (Participants) | 293 | 291
  fHbp (M14459) | 14.7 [10.8 to 19.3] | 21.0 [16.4 to 26.1]
  NadA (96217): number analyzed (Participants) | 293 | 292
  NadA (96217) | 68.9 [63.3 to 74.2] | 78.4 [73.3 to 83.0]
  PorA (NZ98/254): number analyzed (Participants) | 293 | 292
  PorA (NZ98/254) | 8.9 [5.9 to 12.7] | 16.4 [12.4 to 21.2]
  NHBA (M13520) | 17.4 [13.2 to 22.2] | 25.3 [20.4 to 30.6]

34. Secondary Outcome: Percentage of Participants With 4-fold Increase in hSBA Titers Relative to Baseline in Both MenB+MenACWY and MenB Groups After the Second rMenB+OMV NZ Vaccination
Description: The immune response to rMenB+OMV NZ vaccine is evaluated by measuring bactericidal activity against each of the N. meningitidis serogroup B test strains (M14459 [fHbp], 96217 [NadA], NZ98/254 [PorA] and M13520 [NHBA]) in terms of the Four-fold increase defined as: - For a pre-vaccination titer <LOD, a post-vaccination titer of >= 4-fold the LOD or >= LLOQ, whichever is greater, - For a pre-vaccination titer >=LOD but <LLOQ, a post vaccination titer of at least 4-fold the LLOQ, - For a pre-vaccination titer >=LLOQ, a post vaccination titer of at least 4-fold the pre-vaccination titer.
Time Frame: At 1 month after the second rMenB+OMV vaccination (i.e at Day 91) relative to baseline (i.e. Day 1)
Population: as for outcome 26
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MenB+MenACWY Group | MenB Group
Number analyzed (Participants) | 273 | 266
Percentage of participants
  fHbp (M14459): number analyzed (Participants) | 273 | 263
  fHbp (M14459) | 57.1 [51.0 to 63.1] | 64.6 [58.5 to 70.4]
  NadA (96217): number analyzed (Participants) | 273 | 265
  NadA (96217) | 96.0 [92.9 to 98.0] | 98.9 [96.7 to 99.8]
  PorA (NZ98/254): number analyzed (Participants) | 272 | 265
  PorA (NZ98/254) | 51.5 [45.4 to 57.5] | 56.6 [50.4 to 62.7]
  NHBA (M13520): number analyzed (Participants) | 272 | 266
  NHBA (M13520) | 55.1 [49.0 to 61.2] | 53.0 [46.8 to 59.1]

35. Secondary Outcome: Percentage of Participants With hSBA Titers >=LLOQ for Each of the Serogroup A, C, W and Y in Both MenB+MenACWY and MenACWY Groups After MenACWY Vaccination
Description: The immune response to MenACWY vaccines is expressed in terms of percentage of participants with hSBA titers >=LLOQ for each of the serogroup Men A, Men C, Men W and Men Y.
Time Frame: At baseline (Day 1) and at one month after the MenACWY vaccination (i.e. Day 31)
Population: as for outcome 26
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MenB+MenACWY Group | MenACWY Group
Number analyzed (Participants) | 295 | 303
Percentage of participants
  Men A, Baseline (Day 1): number analyzed (Participants) | 267 | 273
  Men A, Baseline (Day 1) | 28.1 [22.8 to 33.9] | 30.0 [24.7 to 35.9]
  Men A, Day 31: number analyzed (Participants) | 290 | 292
  Men A, Day 31 | 99.7 [98.1 to 100] | 99.3 [97.5 to 99.9]
  Men C, Baseline (Day 1): number analyzed (Participants) | 294 | 297
  Men C, Baseline (Day 1) | 46.3 [40.5 to 52.1] | 44.4 [38.7 to 50.3]
  Men C, Day 31: number analyzed (Participants) | 295 | 302
  Men C, Day 31 | 99.0 [97.1 to 99.8] | 98.7 [96.6 to 99.6]
  Men W, Baseline (Day 1): number analyzed (Participants) | 292 | 292
  Men W, Baseline (Day 1) | 27.4 [22.4 to 32.9] | 28.4 [23.3 to 34.0]
  Men W, Day 31 | 100 [98.8 to 100] | 100 [98.8 to 100]
  Men Y, Baseline (Day 1): number analyzed (Participants) | 291 | 296
  Men Y, Baseline (Day 1) | 23.4 [18.6 to 28.7] | 23.0 [18.3 to 28.2]
  Men Y, Day 31 | 99.7 [98.1 to 100] | 99.7 [98.2 to 100]

36. Secondary Outcome: GMRs Against Each of the N. Meningitidis Serogroup Men A, Men C, Men W and Men Y in Both MenB+MenACWY and MenACWY Groups After MenACWY Vaccination
Description: Immune response to MenACWY given with or without rMenB+OMV NZ was measured by bactericidal activity against the four serogroups Men A, Men C, Men W and Men Y in terms of GMRs at one month after MenACWY vaccination compared to the baseline at Day 1/Month 0. GMR was measured within-group.
Time Frame: At 1 month after MenACWY vaccination (i.e.at Day 31) compared to the baseline (Day 1)
Population: as for outcome 26
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | MenB+MenACWY Group | MenACWY Group
Number analyzed (Participants) | 295 | 303
Ratio
  Men A: number analyzed (Participants) | 290 | 292
  Men A | 150.2 [120.1 to 187.8] | 145.0 [115.4 to 182.2]
  Men C: number analyzed (Participants) | 295 | 302
  Men C | 130.0 [97.7 to 173.1] | 131.9 [98.8 to 176.1]
  Men W | 294.2 [229.0 to 378.1] | 279.3 [216.6 to 360.1]
  Men Y | 324.3 [252.2 to 417.0] | 300.0 [232.9 to 386.4]

37. Secondary Outcome: Percentage of Participants With 4-fold Increase in hSBA Titers Against Each of the N. Meningitidis Serogroup Men A, Men C, Men W and Men Y Relative to Baseline in Both MenB+MenACWY and MenACWY Groups After MenACWY Vaccination
Description: The immune response to MenACWY vaccine is evaluated by measuring percentage of participants with 4-fold increase for the four serogroups Men A, Men C, Men W and Men Y. The Four-fold increase defined as: - For a pre-vaccination titer <LOD, a post-vaccination titer of >= 4-fold the LOD or >= LLOQ, whichever is greater, - For a pre-vaccination titer >=LOD but <LLOQ, a post vaccination titer of at least 4-fold the LLOQ, - For a pre-vaccination titer >= LLOQ, a post vaccination titer of at least 4-fold the pre-vaccination titer
Time Frame: At 1 month after MenACWY vaccination (i.e at Day 31) relative to baseline (i.e. Day 1)
Population: as for outcome 26
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MenB+MenACWY Group | MenACWY Group
Number analyzed (Participants) | 293 | 296
Percentage of participants
  Men A: number analyzed (Participants) | 262 | 262
  Men A | 98.5 [96.1 to 99.6] | 98.1 [95.6 to 99.4]
  Men C | 95.2 [92.1 to 97.4] | 95.6 [92.6 to 97.6]
  Men W: number analyzed (Participants) | 291 | 292
  Men W | 98.6 [96.5 to 99.6] | 97.9 [95.6 to 99.2]
  Men Y: number analyzed (Participants) | 290 | 296
  Men Y | 98.6 [96.5 to 99.6] | 98.3 [96.1 to 99.4]

ADVERSE EVENTS:
Time Frame: Solicited AEs: collected during the 7-day follow-up after each vaccination Unsolicited AEs: collected during the 30-day follow-up after each vaccination All-cause mortality, SAEs, MAAEs, AEs leading to withdrawal, and AESIs: - For participants not reaching Day 271 by Protocol Amendment 7: from the first vaccination (Day 1) to Day 271 - For participants past Day 271 by the amendment: from the first vaccination (Day 1) to Day 451
Arm/Group | MenB+MenACWY Group | MenB Group | MenACWY Group
All-Cause Mortality (participants affected / at risk) | 0/310 | 0/308 | 0/320
Serious Adverse Events (participants affected / at risk) | 2/310 | 4/308 | 7/320
Other Adverse Events (participants affected / at risk) | 293/310 | 293/308 | 289/320
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MenB+MenACWY Group (N=310) | MenB Group (N=308) | MenACWY Group (N=320)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1)
Adjustment disorder with depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Drug abuse (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Major depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MenB+MenACWY Group (N=310) | MenB Group (N=308) | MenACWY Group (N=320)
Lymphadenopathy (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Os trigonum (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 3 (3)
Eustachian tube dysfunction (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1)
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Polycystic ovarian syndrome (Endocrine disorders) | 0 (0) | 1 (1) | 1 (1)
Astigmatism (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Episcleritis (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Myopia (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 4 (5) | 5 (5)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 4 (6)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 74 (105) | 90 (119) | 94 (132)
Salivary gland mucocoele (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Tooth impacted (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Toothache (Gastrointestinal disorders) | 5 (5) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (4) | 3 (3) | 6 (6)
Administration site erythema (General disorders) | 28 (39) | 31 (37) | 28 (30)
Administration site induration (General disorders) | 31 (46) | 35 (56) | 25 (33)
Administration site pain (General disorders) | 281 (589) | 282 (597) | 268 (629)
Administration site swelling (General disorders) | 31 (38) | 32 (44) | 26 (33)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 1 (1)
Chills (General disorders) | 2 (2) | 2 (3) | 3 (3)
Fatigue (General disorders) | 152 (265) | 160 (306) | 159 (303)
Feeling of body temperature change (General disorders) | 0 (0) | 0 (0) | 1 (1)
Induration (General disorders) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 1 (1) | 2 (2) | 0 (0)
Injection site bruising (General disorders) | 3 (3) | 1 (2) | 0 (0)
Injection site hypoaesthesia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 1 (1) | 1 (1) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 1 (1) | 0 (0) | 1 (1)
Injection site swelling (General disorders) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 2 (2) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 14 (17) | 23 (26) | 19 (21)
Swelling (General disorders) | 0 (0) | 1 (1) | 1 (1)
Vaccination site bruising (General disorders) | 0 (0) | 1 (1) | 0 (0)
Vaccination site erythema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Vaccination site rash (General disorders) | 1 (1) | 0 (0) | 0 (0)
Vaccination site swelling (General disorders) | 0 (0) | 0 (0) | 1 (1)
Multiple allergies (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Acute sinusitis (Infections and infestations) | 0 (0) | 3 (3) | 3 (3)
Bacterial vaginosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bacterial vulvovaginitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Beta haemolytic streptococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bronchitis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 9 (9) | 5 (5) | 9 (9)
Chlamydial infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Conjunctivitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Fungal infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Gonorrhoea (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Impetigo (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 4 (4) | 10 (10) | 2 (2)
Nasopharyngitis (Infections and infestations) | 11 (11) | 4 (5) | 18 (18)
Otitis externa (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Otitis media acute (Infections and infestations) | 3 (3) | 2 (3) | 1 (1)
Pharyngitis (Infections and infestations) | 2 (2) | 3 (3) | 4 (4)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 3 (3) | 2 (2)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pilonidal disease (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pyuria (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1) | 2 (3) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Sinusitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Stitch abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 4 (5) | 1 (1) | 10 (10)
Urethritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Viral infection (Infections and infestations) | 3 (3) | 3 (3) | 0 (0)
Viral pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
Abdominal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Breast procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 2 (2) | 3 (3) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 3 (3)
Distal clavicular osteolysis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Eye injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Face injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Ligament injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 3 (3)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 4 (5) | 0 (0)
Lip injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Open globe injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 1 (1)
Scar (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Suture related complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Torus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Arthroscopy (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 53 (65) | 46 (66) | 58 (77)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2)
Bone swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Medial tibial stress syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 73 (86) | 81 (112) | 88 (116)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 2 (2)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Tendon pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 3 (3) | 2 (2)
Headache (Nervous system disorders) | 178 (320) | 185 (317) | 185 (345)
Migraine (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 2 (2) | 2 (2) | 1 (1)
Generalised anxiety disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Intentional self-injury (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 3 (3)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Abnormal uterine bleeding (Reproductive system and breast disorders) | 2 (2) | 2 (2) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 5 (7) | 2 (2) | 5 (5)
Gynaecomastia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Varicocele (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 8 (8)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 3 (3) | 5 (5)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 11 (11) | 10 (10)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory symptom (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 3 (3)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hirsutism (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Sensitive skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Pallor (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-10-14): https://cdn.clinicaltrials.gov/large-docs/48/NCT04318548/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-03): https://cdn.clinicaltrials.gov/large-docs/48/NCT04318548/SAP_001.pdf